CLINICAL TRIAL: NCT03488082
Title: Coupling Between Saccadic Adaptation and Visuospatial Perception Process: MRI Study in Humans
Brief Title: MRI Study of Saccadic Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0200; 2018-A00932-53 (Other: ID-RCB)
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: saccadic adaptation; visual-spatial perception; fMRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Measurement of the bold signal (Experimental)
  Interventions: Behavioral: fMRI

INTERVENTIONS:
Behavioral: fMRI — saccadic adaptation (target presentations, with or without target jump) during fMRI exam

SUMMARY:
Accurate execution of our directed behaviors in the immediate environment allows the vast majority of our daily activities. Through the movements of our eyes and different parts of our body, we perceive, explore and act on our environment and can exchange and communicate with others. The mechanisms of sensorimotor adaptation of saccades (saccadic adaptation) contribute on the one hand to maintain the accuracy of saccades in the short, medium and long term, by opposing the deleterious effects of various physiological changes (development, aging), pathological or environmental (optical corrections).

The aim of this study is to identify neuronal structures and networks involved in saccadic adaptation through the study of brain metabolic activation (BOLD) during the development of the adaptation of reactive saccades. The study will be organized in a single session with 3 runs. Each run include 4 blocks: 3 include the double-step target paradigm RND, U+, U-) and one without target jump (STA). The 'U+'/ 'U-'blocks include saccadic trials with forward/backward displacement of the target during a targeting saccade, the 'RND' block include saccadic trials with random target jump (forward or backward) and the 'STA' block are trials without displacement of the target. Each subject will make 12 repetitions of the 4 blocks.

ELIGIBILITY:
Inclusion Criteria:

- Age: 18 to 40 years included,

Exclusion Criteria:

* Known ophthalmological or neurological pathology,
* Non-stabilized medical condition,
* Taking psychotropic treatment,
* No fluency in reading in French,
* Pregnant and / or breastfeeding woman

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
BOLD signal | throughout the behavioral experiment at Day 1
  cerebral activations with fMRI measures when the subject fixates or shifts gaze toward visual targets (behavioral tasks).

SECONDARY OUTCOMES:
Eye movements | during the development of saccadic adaptation (throughout the behavioral experiments at Day 1)
  measurement of the eye movements (saccades) of the subject while fixating and shifting gaze toward visual targets (behavioral tasks).

CONTACTS AND LOCATIONS:
Overall Officials: Denis PELISSON, Principal Investigator — INSERM U1208
Locations (1):
- Inserm U1208, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metais C, Nicolas J, Diarra M, Cheviet A, Koun E, Pelisson D. Neural substrates of saccadic adaptation: Plastic changes versus error processing and forward versus backward learning. Neuroimage. 2022 Nov 15;262:119556. doi: 10.1016/j.neuroimage.2022.119556. Epub 2022 Aug 12. PMID 35964865